CLINICAL TRIAL: NCT00332800
Title: What Impact Does Intensive Vs. Standard Nutritional Supplementary Treatment of Undernourished Stroke Patient Have on Functional Outcome Measures on an Acute Rehabilitation Unit - a Pilot Study
Brief Title: Study Impact of Nutritional Supplementary Treatment of Undernourished Stroke Patient on Functional Outcome Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burke Rehabilitation Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BRC-343
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2006-06-02 (Estimated); Status verified 2005-06

CONDITIONS: Stroke
Keywords: Stroke-Nutritional Supplementation-Functional Recovery
MeSH Terms: conditions — Stroke | interventions — Dietary Supplements

INTERVENTIONS:
Drug: Nutritional Supplementation

SUMMARY:
Undernutrition after stroke is frequent and is due to cognitive impairment, visuospatial perceptive deficits, hemiparesis, depression and dysphagia. The impact of intensive nutritional supplementation on functional outcome measures in undernourished stroke patient has not been studied.

DETAILED DESCRIPTION:
The World Health Organization defines malnutrition as "the cellular imbalance between supply of nutrients and energy and the body's demand for them to ensure growth, maintenance, and specific functions". The prevalence of malnutrition in acute stroke patients varies from 8%- 34%. It has been showed that after an acute stroke malnutrition was present in 16.3% patients on hospital admission, which increased to 26.4% after one week and 35% after two weeks of hospitalization. They also showed that 41% of malnourished stroke patients had poor outcome, based on the presence of urinary or respiratory infection, pressure sores, increased mortality rates, greater neurological deficit and longer length of stay, compared to 14% of malnourished patients who had a better outcome3. Prevalence studies of malnutrition in stroke patients admitted to an acute rehabilitation hospital has varied from 49% to 60%. This high prevalence of undernutrition in post stroke patients is due to: inadequate intake, poor nutritional status prior to their stroke onset, age, immobility with increased muscle wasting, high level of dependency, increased energy demands during the recovery period, depression, and dysphagia. In dysphagic stroke patients this is due to impaired chewing and swallowing from bulbar muscle weakness, and decreased sensation during mastication with oral accumulation of solid food resulting in inadequate nutrient intake. Cognitive, perceptual, visual field deficits and motor apraxia all do contribute to impaired self feeding ability and consequently increase the risk for undernutrition in this population.

Undernutrition has been identified as the most modifiable factor associated with poor functional outcome and increase length of stay. Potter et al in a systematic review of nutritional supplementation in adults suggested that routine nutritional supplementation improved weight and anthropometry, both of which are validated measures of nutritional status; as well as improved functional outcomes. Oral sip feedings has been shown to improve nutritional intake in non-dysphagic patients and improve clinical outcome. Potter et al, in their trial of 381 poorly nourished patients found that high energy and protein oral supplements administered as a medication pass was associated with significantly better energy intake and weight gain, along with a reduction in mortality and an improvement in functional outcome. Thus increased energy and protein is justified in acute post stroke nutritionally compromised patients to improve outcome and decrease mortality.

Oral nutritional supplements have the advantage of the ease of administration irrespective of oral or enteral feeding route, aseptic packaging ensuring patient safety, ability to be administered in different consistencies, reproducibility due to pre-measured formulas, and are established products approved as part of hospital formulary.

Undernutrition assessment and treatment after an acute stroke remains a problem in the hospital setting. We therefore decided to: 1) evaluate what impact aggressive nutritional supplementation in addition to their intake of regular diet has on functional outcome measures; and 2) is there an association between dysphagia and nutritional status post-stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Hemorrhagic and ischemic stroke documented clinically and by neuroimaging.
2. Admission to the Stroke Rehabilitation Service of the Burke Rehabilitation Hospital within 4 weeks of the acute neurological insult.
3. Informed consent, from patient or other responsible person according to Burke IRB standards.
4. Stable medical condition, including cardiac status.
5. Patient able to take diet and medication either orally or via the PEG tube.

Exclusion Criteria:

1. Patients with prior documented history of alcohol abuse, renal and liver diseases, and malabsorption.
2. Patients medically unstable.
3. Patient's terminal ill (e.g., patients with stroke as a complication of a terminal cancer).
4. Patients participating in any other structured therapeutic trial in the acute care hospital or at Burke.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-10; Study Completion 2005-12

PRIMARY OUTCOMES:
Change in total Functional Independence Measure (TFIM) score, and change in the FIM-cognitive and FIm-motor subscores.

SECONDARY OUTCOMES:
Length of stay (LOS)and discharge disposition.

CONTACTS AND LOCATIONS:
Overall Officials: Meheroz H Rabadi, MD, MRCPI, Principal Investigator — Burke Rehabilitation Hospital
Locations (1):
- Burke Rehabilitation Hospital, White Plains, New York, United States